CLINICAL TRIAL: NCT00032331
Title: 18/F-FLUORODEOXYGLUCOSE (FDG) POSITRON EMISSION TOMOGRAPHY (PET) IMAGING IN THE MANAGEMENT OF PATIENTS WITH SOLITARY PULMONARY NODULES
Brief Title: (PET) Imaging in the Management of Patients With Solitary Pulmonary Nodules
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 27
Record Dates: First submitted 2002-03-18; First posted 2002-03-19 (Estimated); Last update posted 2009-01-21 (Estimated); Status verified 2004-01

CONDITIONS: Benign and Malignant Solitary Pulmonary Nodules
Keywords: PET imaging, benign and malignant solitary pulmonary nodules
MeSH Terms: interventions — Magnetic Resonance Spectroscopy

INTERVENTIONS:
Procedure: PET Imaging
Procedure: CT scan

SUMMARY:
All patients with a new, untreated solitary pulmonary nodule (SPN) between 7 mm and 3 cm in diameter identified by chest x-ray, will be approached to undergo positron emission tomography (PET) and computerized tomography (CT). The PET and CT scans will be interpreted independently.

The Primary Care Physician will be provided the results of the baseline chest x-ray and the CT scan, and will be asked for a management and treatment decision. Then the results of the PET will be provided to the Primary Care Physician who will be asked for a management and treatment decision based on all findings (chest x-ray, CT, and PET).

DETAILED DESCRIPTION:
Intervention: All patients will undergo a CT scan and PET imaging. Primary Hypothesis: FDG-PET will be more accurate than existing anatomic modalities (chest x-ray and CT scan) in distinguishing between benign and malignant solitary pulmonary nodules (SPN)? This should expedite the removal of any potentially surgically curable malignant lesion and minimize the number of benign masses and surgically incurable lung neoplasms for which unnecessary thoracotomy is done. Secondary Hypothesis: What is the impact of the results of FDG-PET on the diagnosis made and treatment rendered by the referring physicians? What is the intra- and inter-reader reliability of FDG-PET? What is the effect of FDG-PET on the cost of early management of SPNs when FDG-PET is included in the management paradigm or substituted for CT?

Primary Outcomes: Benign or malignant solitary pulmonary nodules, and their treatment.

Study Abstract: All patients with a new, untreated solitary pulmonary nodule (SPN) between 7 mm and 3 cm in diameter identified by chest x-ray, will be approached to participate in the study. Patients will undergo positron emission tomography (PET) and computerized tomography (CT). The PET and CT scans will be interpreted independently.

The Primary Care Physician will be provided the results of the baseline chest x-ray and the CT scan, and will be asked for a management and treatment decision. Then the results of the PET will be provided to the Primary Care Physician who will be asked for a management and treatment decision based on all findings (chest x-ray, CT, and PET).

Site readers will perform an overview of the CT and PET interpretations and provide a diagnosis of the SPN. There will be an Independent Research Readers Panel which will perform an overview of the CT and PET interpretations and provide a diagnosis of the SPN. These readings will determine inter-reader reliability, and those by the Independent Research Readers Panel will be used as the primary diagnostic measure for the sensitivity and specificity analysis.

The CT and PET diagnoses will be compared with the 'gold standard' (tissue diagnosis, either by fine needle biopsy or surgical pathology, or two year follow-up for changes in the SPN on chest x-ray) to construct Receiver Operating Characteristics (ROC) curves.

There are two substudies - one investigating the economic analysis and one investigating the accuracy of coincidence PET scanning.

ELIGIBILITY:
All patients with a new, untreated solitary pulmonary nodule (SPN) between 7 mm and 3 cm in diameter identified by chest x-ray, will be approached to participate in the study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 500
Dates: Start 1999-01; Study Completion 2003-06